CLINICAL TRIAL: NCT05719441
Title: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial of Combination HIV-Specific Broadly Neutralizing Monoclonal Antibodies Combined With ART Initiation During Acute HIV Infection to Induce HIV Remission
Brief Title: A Clinical Trial of Combination HIV-Specific Broadly Neutralizing Monoclonal Antibodies Combined With ART Initiation During Acute HIV Infection to Induce HIV Remission
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5388; 38662 (Other: DAIDS-ES ID)
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acute HIV Infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: VRC07-523LS + PGT121.414.LS + ART (Experimental)
  Interventions: Biological: VRC07-523LS; Biological: PGT121.414.LS; Drug: ART
- Arm 2: Placebo + ART (Placebo Comparator)
  Interventions: Other: Placebo; Drug: ART

INTERVENTIONS:
Biological: VRC07-523LS — 10 mg/kg intravenous infusion over approximately 15 to 30 minutes once at entry
  Other Names: VRC-HIVMAB075-00-AB
  Arms: Arm 1: VRC07-523LS + PGT121.414.LS + ART
Biological: PGT121.414.LS — 5 mg/kg intravenous infusion over approximately 30 to 60 minutes once at entry
  Other Names: VRC-HIVMAB0107-00-AB
  Arms: Arm 1: VRC07-523LS + PGT121.414.LS + ART
Other: Placebo — Sodium Chloride for Injection USP, 0.9%
  Arms: Arm 2: Placebo + ART
Drug: ART — Bictegravir 50 mg/emtricitabine 200 mg/tenofovir alafenamide 25 mg tablet orally once daily with or without food
  Other Names: Biktarvy

SUMMARY:
A5388 is a phase II, two-arm, randomized, double-blind, placebo-controlled study that will enroll 48 antiretroviral therapy (ART)-naïve adults with acute HIV infection (AHI) in order to determine whether:

* Administration of combination HIV-specific broadly neutralizing antibody (bNAb) therapy in addition to ART during acute HIV infection (AHI) will be safe.
* Participants who receive combination bNAb therapy in addition to ART during AHI will be more likely to demonstrate a delay in time to HIV-1 RNA ≥1,000 copies/mL for 4 consecutive weeks compared to participants who receive placebo plus ART.
* Participants who receive combination bNAb therapy in addition to ART during AHI will demonstrate lower viral reservoirs and enhanced HIV-specific immunity compared to participants who receive placebo plus ART.

ELIGIBILITY:
Inclusion Criteria:

Step 1:

1. Appropriate documentation from medical records of diagnosis of AHI prior to enrollment that includes one of the following:

   1. A detectable HIV-1 RNA within 28 days prior to study entry AND a non-reactive HIV-1 antibody within 7 days prior to entry; OR
   2. A detectable HIV-1 RNA or a reactive HIV-1 antibody within 28 days prior to study entry AND a negative/indeterminate Western Blot (WB) or negative/indeterminate Geenius HIV-1/HIV-2 Supplemental Assay within 7 days prior to entry; OR
   3. A documented non-reactive HIV-1 antibody or negative HIV-1 RNA within 90 days prior to study entry AND a documented reactive HIV-1 antibody or positive WB that is negative for p31 band or a positive Geenius HIV-1/HIV-2 Supplemental Assay that is negative for p31 band within 7 days prior to entry; OR
   4. ARCHITECT or GSCOMBO S/CO ≥10 within 7 days prior to entry AND a non-reactive HIV-1 antibody within 7 days prior to entry; OR
   5. ARCHITECT or GSCOMBO S/CO ≥1 within 7 days prior to entry AND a non-reactive HIV-1 antibody within 7 days prior to entry AND a known prior S/CO <0.5 within 90 days prior to entry; OR
   6. ARCHITECT or GSCOMBO S/CO >0.5 but <10 within 7 days prior to entry AND a non-reactive HIV-1 antibody within 7 days prior to entry AND detectable HIV-1 RNA within 7 days prior to entry
2. The following laboratory values obtained within 21 days prior to entry:

   * Absolute neutrophil count (ANC) ˃1,000/mm3
   * Hemoglobin:

     * >10 g/dL for cisgender men and transgender women
     * >9 g/dL for cisgender women and transgender men
   * Platelet count ˃100,000/mm3
   * Estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation, with consideration for lower rates in special circumstances.
   * ALT (SGPT) ≤2.5 x ULN
   * AST (SGOT) ≤2.5 x ULN
   * Total bilirubin <1.5 x ULN
3. For persons who are able to become pregnant, negative urine or serum pregnancy test within 24 hours prior to study entry.
4. Persons who are able to become pregnant must agree to use two methods of contraception throughout Step 1 if participating in sexual activity that could lead to pregnancy. One contraceptive method must be a highly effective method and the second method of contraception must be a barrier method.
5. Participants of reproductive potential who engage in sexual activity that could lead to their partner's becoming pregnant must agree to use a barrier method of contraception throughout Step 1.
6. Ability and willingness to use a barrier method or abstinence from sexual intercourse with all partners who are vulnerable to HIV or whose HIV serostatus is unknown in order to prevent HIV transmission during Step 2, Step 3, and until plasma HIV-1 RNA is less than the limit of detection after ART restart in Step 4.
7. Age ≥18 and ≤70 years.
8. Ability and willingness to initiate ART at enrollment.
9. Ability and willingness to participate in scheduled study visits, including during the ATI, per Schedule of Evaluations (SOE).
10. Ability and willingness of participant to provide informed consent.

Step 2:

1. Documented negative hepatitis B virus (HBV) surface antigen (HBsAg) obtained within 16 weeks prior to Step 2 registration.
2. Documented negative hepatitis C virus (HCV) antibody (anti-HCV) or negative HCV RNA PCR obtained within 16 weeks prior to Step 2 registration.
3. Receipt of full doses of study infusions at enrollment (VRC07-523LS + PGT121.414.LS or placebo [Sodium Chloride for Injection USP, 0.9%]).
4. HIV-1 RNA <200 copies/mL obtained within 6 weeks prior to Step 2 registration.
5. CD4+ T-cell count ≥450 cells/mm3 obtained within 6 weeks prior to Step 2 registration.
6. For participants who are able to become pregnant, negative serum or urine pregnancy test within 48 hours prior to Step 2 entry.
7. To avoid pregnancy, participants who are able to become pregnant must agree to use contraception or practice abstinence from sexual activity that could lead to pregnancy throughout Step 2.
8. Ability and willingness to use a barrier method or abstinence from sexual intercourse with partners who are vulnerable to HIV or whose HIV serostatus is unknown in order to prevent HIV transmission throughout Step 2.
9. Ability and willingness to interrupt ART.
10. Completion of Step 1.

Step 3:

1. Has not met ART restart criteria.
2. Completion of Step 2.
3. Willing to continue ATI.
4. To avoid pregnancy, participants who are able to become pregnant must agree to use contraception or practice abstinence from sexual activity that could lead to pregnancy throughout Step 3.
5. Ability and willingness to use a barrier method or abstinence from sexual intercourse with all partners who are vulnerable to HIV or whose HIV serostatus is unknown in order to prevent HIV transmission throughout Step 3.

Step 4:

1. Has met any of the ART restart criteria during Step 2 or Step 3. -OR- Has completed Step 3 and is not enrolling to ACTG A5385.
2. To avoid pregnancy, participants who are able to become pregnant must agree to use contraception or practice abstinence from sexual activity that could lead to pregnancy throughout Step 4.
3. Ability and willingness to use a barrier method or abstinence from sexual intercourse with all partners who are vulnerable to HIV or whose HIV serostatus is unknown in order to prevent HIV transmission until plasma HIV-1 RNA is less than the limit of detection after ART restart.

Exclusion Criteria:

Step 1:

1. Previous receipt of immunoglobulin (IgG) therapy.
2. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational (other than for the prevention and/or treatment of SARS-CoV-2/COVID-19).
3. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis in the 2 years prior to enrollment.
4. History of chronic urticaria requiring daily treatment.
5. Receipt of investigational study agent within 28 days prior to enrollment.
6. Past participation in an investigational study of a candidate HIV vaccine or immune prophylaxis for HIV-1 infection with receipt of active product or with receipt of active product or placebo and remains blinded to what they actually received.
7. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months.
8. Use of any immunomodulatory medications within 6 months of study entry including systemic corticosteroids (long-term), immunosuppressants, anti-cancer, interleukins, systemic interferons, systemic chemotherapy, or other medications that the site investigator feels could have an immune modulatory effect.
9. Use of ART for any reason, including pre- or post-exposure prophylaxis, within 60 days prior to study entry.
10. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
11. Known history of active Hepatitis B or Hepatitis C infection.
12. Any acute, chronic, or recent and clinically significant medical condition that, in the opinion of the site investigator, would interfere with adherence to study requirements or jeopardize the safety or rights of the participant.
13. History of or current clinical atherosclerotic cardiovascular disease (ASCVD) as defined by 2013 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines, including a previous diagnosis of any of the following:

    * Acute myocardial infarction
    * Acute coronary syndromes
    * Stable or unstable angina
    * Coronary or other arterial revascularization
    * Stroke
    * TIA
    * Peripheral arterial disease presumed to be of atherosclerotic origin
14. Currently breastfeeding or pregnant.
15. Weight >115 kg.
16. Use of prohibited medications for bictegravir, emtricitabine, and tenofovir alafenamide (refer to protocol section 5.8) within 7 days prior to entry, or planned use of prohibited medications during the period of study participation.
17. Absence of adequate venous access for the administration of infusion or for phlebotomy to assess for the primary study endpoint.

Step 2:

1. Viral failure, as defined in protocol section 6.2.4, after Step 1 week 24.
2. Failure to initiate ART in Step 1.
3. Receipt of any non-nucleoside reverse transcriptase inhibitor (NNRTI) or long-acting ART (any therapy dosed at an interval less than daily), such as cabotegravir or rilpivirine injections, after Step 1 entry.
4. Receipt of any immunoglobulin therapy or immunomodulatory medications after Step 1 entry including systemic corticosteroids (long-term), immunosuppressants, anti-cancer, interleukins, systemic interferons, systemic chemotherapy, or other medications that the site investigator feels could have an immune modulatory effect.
5. Does not have HIV-1.
6. Participant was in Fiebig stage VI at the time of study entry.
7. Failure by the participant to attend three consecutive Step 1 study visits.
8. Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during ATI.
9. Pregnancy or breastfeeding.
10. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Step 3:

1. Transfer to A5385 (The Post-Intervention Cohort Study).
2. ART restart in Step 2.
3. Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during analytic treatment interruption.
4. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Step 4:

1. Unwillingness or inability to restart ART after meeting an ART restart criterion in Step 2 or Step 3.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2028-04-06 (Estimated); Study Completion 2028-09-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade ≥2 AE or SAE that are possibly, probably, or definitely related to the study bNAbs during Step 1 | Week 0 to end of Step 1
Time from ART discontinuation to HIV-1 RNA ≥1,000 copies/mL for 4 consecutive weeks during Step 2 | From Step 2 entry through 24 weeks after ART interruption

SECONDARY OUTCOMES:
Time from ART discontinuation to first documented HIV-1 RNA viral rebound of ≥50 copies/mL during Step 2 | From Step 2 entry through 24 weeks after ART interruption
Time from ART discontinuation to first documented HIV-1 RNA viral rebound of ≥200 copies/mL during Step 2 | From Step 2 entry through 24 weeks after ART interruption
Time from ART discontinuation to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL during Step 2 | From Step 2 entry through 24 weeks after ART interruption
Proportion of study participants who undergo ATI with HIV-1 RNA <200 copies/mL at 24 weeks after ART interruption, without indication of ART restart | From Step 2 entry through 24 weeks after ART interruption
Time from ART discontinuation to ART restart for an HIV-related reason (virologic, immunologic and clinical criteria) during Step 2 | From Step 2 entry through 24 weeks after ART interruption
Frequency of participants maintained off ART at each visit during Step 2 | From Step 2 entry through 24 weeks after ART interruption
Change in CD4+/CD8+ T-cell counts during Step 2 | From Step 2 entry through 24 weeks after ART interruption
Area under the curve (AUC) of VRC07-523LS and PGT121.414.LS when administered together | Week 0 to end of Step 3
Half-life of VRC07-523LS and PGT121.414.LS when administered together | Week 0 to end of Step 3
Cmax of VRC07-523LS and PGT121.414.LS when administered together | Week 0 to end of Step 3
Cmin of VRC07-523LS and PGT121.414.LS when administered together | Week 0 to end of Step 3
Clearance (Cl/F) of VRC07-523LS and PGT121.414.LS when administered together | Week 0 to end of Step 3
Volume of distribution of VRC07-523LS and PGT121.414.LS when administered together | Week 0 to end of Step 3

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Crowell, MD, PhD, Study Chair — U.S. Military HIV Research Program CTU
Locations (36):
- United States (32):
  - 31788, Alabama CRS, Birmingham, Alabama
  - 1201, University of Southern California CRS, Los Angeles, California
  - 601, University of California, Los Angeles CARE Center CRS, Los Angeles, California
  - 701, UCSD Antiviral Research Center CRS, San Diego, California
  - 801, University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - 603, Harbor University of California Los Angeles Center CRS, Torrance, California
  - 6101, University of Colorado Hospital CRS, Aurora, Colorado
  - 31791, Whitman-Walker Institute, Inc. CRS, Washington D.C., District of Columbia
  - 5802, The Ponce de Leon Center CRS, Atlanta, Georgia
  - 2701, Northwestern University CRS, Chicago, Illinois
  - 2702, Rush University CRS, Chicago, Illinois
  - 201, Johns Hopkins University CRS, Baltimore, Maryland
  - 101, Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - 107, Brigham and Women's Hospital Therapeutics (BWH TCRS) CRS, Boston, Massachusetts
  - 2101, Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - 31786, New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - 7804, Weill Cornell Chelsea CRS, New York, New York
  - 30329, Columbia Physicians & Surgeons (P&S) CRS, New York, New York
  - 7803, Weill Cornell Uptown CRS, New York, New York
  - 31787, University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - 3201, Chapel Hill CRS, Chapel Hill, North Carolina
  - 3203, Greensboro CRS, Greensboro, North Carolina
  - 2401, Cincinnati CRS, Cincinnati, Ohio
  - 2501, Case CRS, Cleveland, Ohio
  - 2301, Ohio State University CRS, Columbus, Ohio
  - 6201, Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - 1001, University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - 2951, The Miriam Hospital (TMH) CRS, Providence, Rhode Island
  - 3652, Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - 31443, Trinity Health and Wellness Center CRS, Dallas, Texas
  - 31473, Houston AIDS Research Team CRS, Houston, Texas
  - 1401, University of Washington Positive Research CRS, Seattle, Washington
- Brazil (2):
  - 12201, Hospital Nossa Senhora da Conceicao CRS, Porto Alegre
  - 12101, Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- Peru (2):
  - 11302, San Miguel CRS, San Miguel, Lima region
  - 11301, Barranco CRS, Lima

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/aboutactg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.